CLINICAL TRIAL: NCT04490967
Title: Topical Silymarin Cream Versus Salicylic Acid Peeling in Treatment of Acne Vulgaris: Split Face Study
Brief Title: Silymarin Cream Versus Salicylic Acid in Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Gamal Ahmed Makhlouf, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMVSA
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Silymarin; Silybin; Salicylic Acid

STUDY DESIGN:
Intervention Model Description: Patients will use salicylic acid 30% peeling on the right side of the face and topical Silymarin 1.4% cream on the left side.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silymarin and salicylic acid (Experimental): There will be one group of patients, that will use salicylic acid peeling on the right side of the face and topical Silymarin cream on the left side
  Interventions: Combination Product: Silymarin; Procedure: Salicylic acid

INTERVENTIONS:
Combination Product: Silymarin — Silymarin 1.4% cream will be used on the left side of the face twice daily (home use).
  Other Names: Silybin, Silybum, Marian thistle.
Procedure: Salicylic acid — Patients will have salicylic acid 30% peeling on the right side of the face as a peeling session every two weeks. Sessions will be done by well trained physician.
  Other Names: 2-hydroxybenzoic acid

SUMMARY:
Acne vulgaris is a disease of the pilosebaceous unit that causes noninflammatory lesions (open and closed comedones), inflammatory lesions (papules, pustules, and nodules), and varying degrees of scarring. Acne vulgaris is an extremely common condition with a lifetime prevalence of approximately 85% and occurs mostly during adolescence.

Acne vulgaris leads to significant morbidity that is associated with residual scarring and psychological disturbances such as poor self-image, depression, and anxiety, which leads to a negative impact on quality of life.

The treatment of acne vulgaris is challenging and often chronic, with high rates of failure and numerous choices. Frequent evaluations (i.e., every 8-12 weeks) are important to enable appropriate monitoring, manage adverse effects, and evaluate for medication compliance.

Topical therapies are considered one of the mainstay treatments for patients with mild-to-moderate acne.

DETAILED DESCRIPTION:
Chemical peeling is one of the most common cosmetic procedures in medical practice and has been used for decades. It is defined as the application of chemical agents, of variable strength, on the skin that results in controlled destruction of the epidermis and dermis. The induced exfoliation is followed by dermal and epidermal regeneration from adjacent epithelium and skin adnexa, which results in improved surface texture and appearance of the skin. This is a simple and cost-effective procedure with several dermatological applications.

Salicylic acid is a 2-hydroxybenzoic acid used for superficial peeling due to its strong keratolytic and comedolytic properties. It promotes shedding of epidermal cells and due to its lipophilic properties can penetrate comedones and pores to prevent clogging and neutralize bacteria. It promotes desquamation of the upper lipophilic layers of the stratum corneum. These chemical properties explain its popularity and success in acne patients. Also, it has well-documented anti-inflammatory properties.

Silymarin is a standardized extract from S. marianum seeds, is traditionally used as a hepatoprotective agent for its potent regenerative properties. Lately, Silymarin is utilized in dermatological and cosmetic preparations for its antioxidant effect anti-inflammatory and immunomodulatory properties.

Various studies have been created to evaluate the efficacy of Silymarin in UV protection, prevention against skin cancer and against actinic keratosis.

Silymarin showed efficacy the treatment of Rosacea, Melasma, Vitiligo, Psoriasis, atopic dermatitis and contact dermatitis . Other studies showed that Silymarin has anti aging properties and potential action for wound healing .

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age.
* Patients with mild and moderate acne vulgaris.
* Patients with Fitzpatrick skin type III, IV and V.

Exclusion Criteria:

* Severe acne.
* Patients under treatment with contraceptive pills or any kind of systemic or topic acne medication (isotretinoin, antibiotics, topical products).
* History of hypertrophic/keloid scar formation.
* Pregnancy.
* Recurrent herpes infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the medication: number of inflammatory, non-inflammatory and total lesions | 12 weeks
  counting the number of inflammatory, non-inflammatory and total lesions at baseline and every 4 weeks during the treatment
assessment of tolerability: interviewing the patients | 12 weeks
  interviewing the patients about any sign/symptom of adverse reactions (erythema, peeling, burning sensation, dryness and pruritus)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bhate K, Williams HC. Epidemiology of acne vulgaris. Br J Dermatol. 2013 Mar;168(3):474-85. doi: 10.1111/bjd.12149. PMID 23210645
- [Background] Ramos-e-Silva M, Ramos-e-Silva S, Carneiro S. Acne in women. Br J Dermatol. 2015 Jul;172 Suppl 1:20-6. doi: 10.1111/bjd.13638. PMID 25597414
- [Background] Kamangar F, Shinkai K. Acne in the adult female patient: a practical approach. Int J Dermatol. 2012 Oct;51(10):1162-74. doi: 10.1111/j.1365-4632.2012.05519.x. PMID 22994662
- [Background] Nast A, Dreno B, Bettoli V, Degitz K, Erdmann R, Finlay AY, Ganceviciene R, Haedersdal M, Layton A, Lopez-Estebaranz JL, Ochsendorf F, Oprica C, Rosumeck S, Rzany B, Sammain A, Simonart T, Veien NK, Zivkovic MV, Zouboulis CC, Gollnick H; European Dermatology Forum. European evidence-based (S3) guidelines for the treatment of acne. J Eur Acad Dermatol Venereol. 2012 Feb;26 Suppl 1:1-29. doi: 10.1111/j.1468-3083.2011.04374.x. No abstract available. PMID 22356611
- [Background] Al-Talib H, Al-Khateeb A, Hameed A, Murugaiah C. Efficacy and safety of superficial chemical peeling in treatment of active acne vulgaris. An Bras Dermatol. 2017 Mar-Apr;92(2):212-216. doi: 10.1590/abd1806-4841.20175273. PMID 28538881
- [Background] Rendon MI, Berson DS, Cohen JL, Roberts WE, Starker I, Wang B. Evidence and considerations in the application of chemical peels in skin disorders and aesthetic resurfacing. J Clin Aesthet Dermatol. 2010 Jul;3(7):32-43. PMID 20725555
- [Background] Clark E, Scerri L. Superficial and medium-depth chemical peels. Clin Dermatol. 2008 Mar-Apr;26(2):209-18. doi: 10.1016/j.clindermatol.2007.09.015. PMID 18472062
- [Background] Arif T. Salicylic acid as a peeling agent: a comprehensive review. Clin Cosmet Investig Dermatol. 2015 Aug 26;8:455-61. doi: 10.2147/CCID.S84765. eCollection 2015. PMID 26347269
- [Background] Lee HS, Kim IH. Salicylic acid peels for the treatment of acne vulgaris in Asian patients. Dermatol Surg. 2003 Dec;29(12):1196-9; discussion 1199. doi: 10.1111/j.1524-4725.2003.29384.x. PMID 14725662
- [Background] Handog EB, Datuin MS, Singzon IA. Chemical peels for acne and acne scars in asians: evidence based review. J Cutan Aesthet Surg. 2012 Oct;5(4):239-46. doi: 10.4103/0974-2077.104911. PMID 23378705
- [Background] Vaid M, Katiyar SK. Molecular mechanisms of inhibition of photocarcinogenesis by silymarin, a phytochemical from milk thistle (Silybum marianum L. Gaertn.) (Review). Int J Oncol. 2010 May;36(5):1053-60. doi: 10.3892/ijo_00000586. PMID 20372777
- [Background] Surai PF. Silymarin as a Natural Antioxidant: An Overview of the Current Evidence and Perspectives. Antioxidants (Basel). 2015 Mar 20;4(1):204-47. doi: 10.3390/antiox4010204. PMID 26785346
- [Background] Katiyar SK, Mantena SK, Meeran SM. Silymarin protects epidermal keratinocytes from ultraviolet radiation-induced apoptosis and DNA damage by nucleotide excision repair mechanism. PLoS One. 2011;6(6):e21410. doi: 10.1371/journal.pone.0021410. Epub 2011 Jun 22. PMID 21731736
- [Background] Meeran SM, Katiyar S, Elmets CA, Katiyar SK. Silymarin inhibits UV radiation-induced immunosuppression through augmentation of interleukin-12 in mice. Mol Cancer Ther. 2006 Jul;5(7):1660-8. doi: 10.1158/1535-7163.MCT-06-0095. PMID 16891451
- [Background] Katiyar SK, Meleth S, Sharma SD. Silymarin, a flavonoid from milk thistle (Silybum marianum L.), inhibits UV-induced oxidative stress through targeting infiltrating CD11b+ cells in mouse skin. Photochem Photobiol. 2008 Mar-Apr;84(2):266-71. doi: 10.1111/j.1751-1097.2007.00241.x. Epub 2007 Nov 28. PMID 18221354
- [Background] Katiyar SK. Treatment of silymarin, a plant flavonoid, prevents ultraviolet light-induced immune suppression and oxidative stress in mouse skin. Int J Oncol. 2002 Dec;21(6):1213-22. PMID 12429970
- [Background] Vaid M, Prasad R, Singh T, Elmets CA, Xu H, Katiyar SK. Silymarin inhibits ultraviolet radiation-induced immune suppression through DNA repair-dependent activation of dendritic cells and stimulation of effector T cells. Biochem Pharmacol. 2013 Apr 15;85(8):1066-76. doi: 10.1016/j.bcp.2013.01.026. Epub 2013 Feb 5. PMID 23395695
- [Background] Vaid M, Prasad R, Sun Q, Katiyar SK. Silymarin targets beta-catenin signaling in blocking migration/invasion of human melanoma cells. PLoS One. 2011;6(7):e23000. doi: 10.1371/journal.pone.0023000. Epub 2011 Jul 28. PMID 21829575 (Retraction: PMID 30596791 PLoS One. 2018 Dec 31;13(12):e0210344)
- [Background] Chatterjee ML, Agarwal R, Mukhtar H. Ultraviolet B radiation-induced DNA lesions in mouse epidermis: an assessment using a novel 32P-postlabelling technique. Biochem Biophys Res Commun. 1996 Dec 13;229(2):590-5. doi: 10.1006/bbrc.1996.1848. PMID 8954942
- [Background] Berman B, Amini S. Pharmacotherapy of actinic keratosis: an update. Expert Opin Pharmacother. 2012 Sep;13(13):1847-71. doi: 10.1517/14656566.2012.716039. PMID 22888917
- [Background] Berardesca E, Cameli N, Cavallotti C, Levy JL, Pierard GE, de Paoli Ambrosi G. Combined effects of silymarin and methylsulfonylmethane in the management of rosacea: clinical and instrumental evaluation. J Cosmet Dermatol. 2008 Mar;7(1):8-14. doi: 10.1111/j.1473-2165.2008.00355.x. PMID 18254805
- [Background] Svobodova A, Zdarilova A, Walterova D, Vostalova J. Flavonolignans from Silybum marianum moderate UVA-induced oxidative damage to HaCaT keratinocytes. J Dermatol Sci. 2007 Dec;48(3):213-24. doi: 10.1016/j.jdermsci.2007.06.008. Epub 2007 Aug 3. PMID 17689055
- [Background] Altaei T. The treatment of melasma by silymarin cream. BMC Dermatol. 2012 Oct 2;12:18. doi: 10.1186/1471-5945-12-18. PMID 23031632
- [Background] Sehgal VN. Role of tacrolimus (FK506) 0.1% ointment WW in vitiligo in children and imperatives of combine therapy with Trioxsalen and Silymarin suspension in progressive vitiligo. J Eur Acad Dermatol Venereol. 2009 Oct;23(10):1218-9. doi: 10.1111/j.1468-3083.2009.03128.x. Epub 2009 Mar 3. No abstract available. PMID 19192018
- [Background] Fiebrich F, Koch H. Silymarin, an inhibitor of lipoxygenase. Experientia. 1979 Dec 15;35(12):1548-60. doi: 10.1007/BF01953184. PMID 118048
- [Background] Koch HP, Bachner J, Loffler E. Silymarin: potent inhibitor of cyclic AMP phosphodiesterase. Methods Find Exp Clin Pharmacol. 1985 Aug;7(8):409-13. PMID 3001454
- [Background] Kang JS, Yoon WK, Han MH, Lee H, Lee CW, Lee KH, Han SB, Lee K, Yang KH, Park SK, Kim HM. Inhibition of atopic dermatitis by topical application of silymarin in NC/Nga mice. Int Immunopharmacol. 2008 Oct;8(10):1475-80. doi: 10.1016/j.intimp.2008.06.004. Epub 2008 Jun 30. PMID 18593606
- [Background] Mady FM, Essa H, El-Ammawi T, Abdelkader H, Hussein AK. Formulation and clinical evaluation of silymarin pluronic-lecithin organogels for treatment of atopic dermatitis. Drug Des Devel Ther. 2016 Mar 10;10:1101-10. doi: 10.2147/DDDT.S103423. eCollection 2016. PMID 27022248
- [Background] Han MH, Yoon WK, Lee H, Han SB, Lee K, Park SK, Yang KH, Kim HM, Kang JS. Topical application of silymarin reduces chemical-induced irritant contact dermatitis in BALB/c mice. Int Immunopharmacol. 2007 Dec 15;7(13):1651-8. doi: 10.1016/j.intimp.2007.08.019. Epub 2007 Sep 14. PMID 17996674
- [Background] Pientaweeratch S, Panapisal V, Tansirikongkol A. Antioxidant, anti-collagenase and anti-elastase activities of Phyllanthus emblica, Manilkara zapota and silymarin: an in vitro comparative study for anti-aging applications. Pharm Biol. 2016 Sep;54(9):1865-72. doi: 10.3109/13880209.2015.1133658. Epub 2016 Feb 24. PMID 26912420
- [Background] Sharifi R, Rastegar H, Kamalinejad M, Dehpour AR, Tavangar SM, Paknejad M, Mehrabani Natanzi M, Ghannadian N, Akbari M, Pasalar P. Effect of topical application of silymarin (Silybum marianum) on excision wound healing in albino rats. Acta Med Iran. 2012;50(9):583-8. PMID 23165806